CLINICAL TRIAL: NCT07355933
Title: Metabolic Flexibility, Eating Behavior and Adipose Tissue Expandability: Role of This Triad in the Propensity to Human Obesity.
Brief Title: Metabolic Flexibility and Metabolic Heath in Human Obesity
Acronym: PROB
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jose Galgani (Other)
Collaborators: Agencia Nacional de Investigación y Desarrollo (Other)
Responsible Party: Sponsor-Investigator, Jose Galgani, Responsible Principal Investigator, Pontificia Universidad Catolica de Chile
Organization: Pontificia Universidad Catolica de Chile (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 200602001
Record Dates: First submitted 2025-07-25; First posted 2026-01-21 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2025-07

CONDITIONS: Obesity
Keywords: OBESITY; WEIGHT LOSS; EATING BEHAVIOR; METABOLIC FLEXIBILITY; BODY COMPOSITION
MeSH Terms: conditions — Obesity; Weight Loss; Feeding Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Weight Loss Intervention (Other): Individuals with overweight or obesity will undergo dietary energy restriction aimed to induce 8 to 12% weight loss after 12 weeks. For 3 to 5 weeks, body weight will be maintained.
  Interventions: Other: Body Weight Loss

INTERVENTIONS:
Other: Body Weight Loss — Individuals will be prescribed a hypocaloric diet (1300 kcal/d). Individuals will receive a booklet detailing the type of meals and foods to be consumed in each mealtime. A dietitian will explain how to enhance dietary compliance. Every two weeks, body weight, vital signs, and adverse events will be monitored. In addition, food recalls will be conducted in order to optimize dietary energy restriction compliance. During weight maintenance, energy intake will be adjusted to energy requirements to maintain weight stability (±2.5 kg) for at least 3 weeks. During weight loss and maintenance, participants will be instructed to maintain their customary physical activity.

SUMMARY:
This observational study explores the relationship between improvements in metabolic health following weight loss and changes in whole-body fat mass and its distribution. The study focuses on adult men and women with excess body weight undergoing dietary energy restriction over 12 weeks. The primary research question is: Does a greater reduction in fat mass for a given weight loss correlate with more significant improvements in metabolic health?

DETAILED DESCRIPTION:
Obesity is a well-established risk factor for disruptions in metabolic health, which often precede cardiovascular disease and type-2 diabetes. While the precise pathophysiological mechanisms linking obesity to these conditions remain unclear, it is widely acknowledged that an increase in fat mass plays a central role, including the expansion of adipose tissue and the accumulation of lipids in non-adipose tissues. As a result, a primary approach to improving metabolic health is to reduce fat mass through negative energy balance. However, lifestyle changes or pharmacological interventions aimed at inducing a negative energy balance do not exclusively target fat mass and often result in the loss of fat-free mass to varying degrees. Given that higher fat mass, rather than fat-free mass, is more strongly associated with impaired metabolic health, strategies that maximize fat mass loss while preserving fat-free mass may offer more significant benefits for metabolic health. Surprisingly, there is a lack of evidence to support this hypothesis. To address this gap, it will be evaluated the relationship between changes in metabolic health and body composition, independent of overall weight loss, in individuals with overweight or obesity undergoing dietary energy restriction. It is hypothesized that greater fat mass reduction will be linked to more substantial improvements in metabolic health for a given weight loss.

ELIGIBILITY:
Inclusion criteria

* males or females
* 30-55 y old
* physically inactive (<600 MET´min/wk of self-reported moderate-vigorous physical activity
* stable body weight for at least the past 6 months (±2 kg)
* healthy according to medical history and routine hematology and biochemistry.

Exclusion criteria

* Individuals with physiological (pregnancy, lactation) or pathological (under drug therapy for and/or having cardiovascular, liver, kidney, thyroid diseases)
* conditions affecting energy metabolism or eating behavior
* Subjects having low-fat (<20% energy) or low-carbohydrate (<45% energy) diets
* Smokers and alcohol abusers

Ages: 30 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 74 (Actual)
Dates: Start 2022-09-23 (Actual); Primary Completion 2025-01-06 (Actual); Study Completion 2025-01-06 (Actual)

PRIMARY OUTCOMES:
Fasting serum triglyceride concentration | From enrollment to the end of weight maintenance period at 15-20 weeks
  In overnight fasted individuals, a blood sample will be drawn. Serum will be isolated and stored at -80C until assessment.

SECONDARY OUTCOMES:
HOMA-IR | From enrollment to the end of weight maintenance period at 15-20 weeks.
  In overnight fasted individuals, a blood sample will be drawn for glucose and insulin assessment. HOMA-IR will be calculated using this formula: (glucose, mM * insulin, uU/mL)/22.5. Serum/Plasma will be isolated and stored at -80C until assessment.

CONTACTS AND LOCATIONS:
Locations (1):
- Avda. Libertador Bernardo O´Higgins 340. Santiago. Chile., Santiago, Santiago Metropolitan, Chile

IPD SHARING:
Plan to Share IPD: No